CLINICAL TRIAL: NCT04372004
Title: Comparison of the Efficacy of Rapid Tests to Identify COVID-19 Infection (CATCh COVID-19)
Acronym: CATCH COVID-19
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Texas Cardiac Arrhythmia Research Foundation (Other)
Responsible Party: Principal Investigator, Andrea Natale, Executive Medical Director, Texas Cardiac Arrhythmia Research Foundation
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: TCAI_CATCH COVID-19
Record Dates: First submitted 2020-04-29; First posted 2020-05-01 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-05

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Diagnostic Tests, Routine

STUDY DESIGN:
Intervention Model Description: Each subject will be tested using 3 different samples on two testing platforms (serology and viral-RNA detection)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Viral RNA test using nasopharyngeal swab (Active Comparator)
  Interventions: Diagnostic Test: diagnostic tests for COVID-19 infection
- Viral RNA test using sputum (Active Comparator)
  Interventions: Diagnostic Test: diagnostic tests for COVID-19 infection
- Serology test using blood (Active Comparator)
  Interventions: Diagnostic Test: diagnostic tests for COVID-19 infection

INTERVENTIONS:
Diagnostic Test: diagnostic tests for COVID-19 infection — Compare the efficacy of diagnostic tests for COVID-19 infection in detecting antibodies and viral-RNA

SUMMARY:
This study is designed to compare the efficacy of detection of COVID-19 infection using the serology test in blood sample and the PCR-based test in the nasopharyngeal (NP) and sputum sample. Furthermore, it aims to evaluate the temporal trend of appearance of IgM and IgG in blood.

DETAILED DESCRIPTION:
The investigators hypothesize that viral-RNA test using sputum will be equally efficient as the test performed in NP swab. Moreover, the serology test and the PCR-based test will be comparable in efficacy for detection of infection

ELIGIBILITY:
Inclusion Criteria:

* • Male or female over 18 years of age at the time of enrollment

  * Current symptoms of COVID-19 ; fever alone or fever and at least one of the following symptoms need to be present

    * Dry cough
    * Sore throat
    * Shortness of breath
    * Chills
    * Muscle pain
    * Headache
    * New loss of taste or smell
    * Chills with repeated shaking

Exclusion Criteria:

* • Unwilling to provide informed consent

  * Unwilling to undergo bi-weekly serological test during the 1-month enrollment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-05-08 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
detection of viral infection using serology and viral-RNA detection kits | 1 day
  Detection of viral infection in the two test platforms using 3 specimen (blood, nasal swab and sputum) from the same subject, in detecting COVID-19 infection

SECONDARY OUTCOMES:
Temporal trend of antibodies in blood | 1 month
  Temporal trend of the IgM and IgG production in response to the infection by conducting serial serology tests at bi-weekly interval

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Cardiac Arrhythmia Institute, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No